CLINICAL TRIAL: NCT02282904
Title: Haploidentical Transplant for Patients With Chronic Granulomatous Disease (CGD) Using Post-Transplant Cyclophosphamide
Brief Title: Haploidentical Transplant for People With Chronic Granulomatous Disease Using Post Transplant Cyclophosphamide
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150007; 15-I-0007 (Other: NIH)
Record Dates: First submitted 2014-11-04; First posted 2014-11-05 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-12-10

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic Granulomatous Disease; Halo-Identical Protocol; Transplant
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Sirolimus; Cyclophosphamide; fludarabine; fludarabine phosphate; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CGD Recipient (Experimental): CGD patients that will undergo haplo transplantation with post-transplant cyclophosphamide as described
  Interventions: Drug: Sirolimus; Biological: Donor peripheral blood stem cells.; Drug: Cyclophosphamide post transplant; Radiation: Total body 200cGy; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Busulfan

INTERVENTIONS:
Drug: Sirolimus — For pediatric patients: Begin sirolimus 1 mg/m2 PO q4h for 3 doses, then 1 mg/m2 once a day (QD). For adult patients, begin sirolimus 5 mg PO q4h for 3 doses, then 5 mg once a day (QD).
  Doses may be adjusted to maintain trough levels between 8-14 ng/ml. Recipients will take sirolimus from Day +5 to at least Day 100 (minimum).
  Other Names: Rapamycin
Biological: Donor peripheral blood stem cells. — Infuse donor graft.
Drug: Cyclophosphamide post transplant — 50 mg/kg/d IV infused over 90 minutes. Day +3 and +4
  Other Names: Cytoxan post transplant
Radiation: Total body 200cGy — Day -1
Drug: Cyclophosphamide — 14.5 mg/kg IV over one hour Day -6 and -5
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m2 over 30 minutes Day -6 through Day -2
  Other Names: Fludara
Drug: Busulfan — Busulfan 3.2 mg/kg IV once daily over 2-3 hours Day -4,-3,-2
  Other Names: Busulfex

SUMMARY:
Background:

- Chronic Granulomatous Disease (CGD) causes immune system problems. Treatment is usually a bone marrow transplant from a fully matched donor. Researchers want to try using partially matched donors for patients who do not have a fully matched donor available. The researchers will also use the drug cyclophosphamide to try to improve the outcomes when using a partially matched donor.

Objective:

- To learn the effectiveness of using cyclophosphamide with a transplant from a partially matched donor in treating CGD.

Eligibility:

- Recipients: age 2-65 with CGD with an ongoing infection that has not been cured by standard treatment and no fully matched donor available in an appropriate timeframe.

Design:

* Recipients will:

  * be admitted to the hospital 2 weeks before transplant.
  * be screened with blood and urine tests, breathing and heart health tests, X-rays, and/or magnetic resonance imaging. They may have a bone marrow aspiration and biopsy.
* meet with a social worker and dentist.
* get chemotherapy, radiation, and other medicines.
* get an intravenous (IV) catheter in their chest.
* have the transplant.
* get more medicines and standard supportive care.
* have blood drawn frequently.
* have to stay in the Washington, D.C. area for 3 months post-transplant.
* be followed closely for the first 6 months, and then less frequently for at least 5 years.

DETAILED DESCRIPTION:
Allogeneic transplant using HLA matched donors, both related and unrelated, has proven curative for patients with various immunodeficiencies, including those with ongoing infections. However donor availability remains a limiting factor in the application of this treatment modality. The use of haploidentical donors has in the past been fraught with a greater rate of complications related to both higher rates of GvHD and delayed immunorecovery. Newer transplant regimens appear to have diminished these risks and improved outcomes. We propose using a subablative conditioning regimen followed by post-transplant cyclophosphamide for patients with CGD who do not have an HLA matched donor but whose circumstances necessitate the use of a potentially curative, albeit high-risk treatment modality.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have sufficient complications from underlying disease to warrant undergoing transplantation
* Ages 2 years - 65 years
* No appropriate HLA matched donor (available donor has greater than 1 mismatch or the single mismatch is not at DQ for unrelated donors (including cord blood products), or no available 6 out of 6 HLA matched related donor), or patients who may have an unrelated donor, but whose clinical status is such that the time required to obtain an unrelated donor would be life threatening.
* HLA haploidentical family donor graft available.
* Ability to comprehend and willingness to sign the informed consent or have a parent/guardian consent if the donor is a minor; assent being obtained from minors as appropriate
* Must be HIV negative
* Must not be pregnant (confirmed by a negative serum beta-human chorionic gonadotropin (Beta-hCG) for women of child-bearing potential) or breastfeeding
* Must be able to stay within one hour s travel of the NIH for the first 3 months after transplantation and have a family member or other designated companion to stay with during the post-transplant period.
* Must provide a durable power of attorney for health care decisions to an appropriate adult relative or guardian in accordance to NIH Form-200 NIH Durable Power of Attorney for Health Care Decision Making.
* Where appropriate, subjects must agree to use contraception for 3 months post-transplant

EXCLUSION CRITERIA:

* Major anticipated illness or organ failure incompatible with survival from Allo-transplant
* Inadequate collection from prospective donors.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10-23; Primary Completion 2019-04-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] Reisner Y, Hagin D, Martelli MF. Haploidentical hematopoietic transplantation: current status and future perspectives. Blood. 2011 Dec 1;118(23):6006-17. doi: 10.1182/blood-2011-07-338822. Epub 2011 Sep 14. PMID 21921045
- [Background] Munchel A, Kesserwan C, Symons HJ, Luznik L, Kasamon YL, Jones RJ, Fuchs EJ. Nonmyeloablative, HLA-haploidentical bone marrow transplantation with high dose, post-transplantation cyclophosphamide. Pediatr Rep. 2011 Jun 22;3 Suppl 2(Suppl 2):e15. doi: 10.4081/pr.2011.s2.e15. PMID 22053277

RESULTS

PARTICIPANT FLOW:
Groups:
- CGD Recipient: CGD patients that will undergo haplo transplantation with post-transplant cyclophosphamide as described
  Sirolimus: For pediatric patients: Begin sirolimus 1 mg/m2 PO q4h for 3 doses, then 1 mg/m2 once a day (QD). For adult patients, begin sirolimus 5 mg PO q4h for 3 doses, then 5 mg once a day (QD).
  Doses may be adjusted to maintain trough levels between 8-14 ng/ml. Recipients will take sirolimus from Day +5 to at least Day 100 (minimum).
  Donor peripheral blood stem cells.: Infuse donor graft.
  Cyclophosphamide post transplant: 50 mg/kg/d IV infused over 90 minutes. Day +3 and +4
  Total body 200cGy: Day -1
  Cyclophosphamide: 14.5 mg/kg IV over one hour Day -6 and -5
  Fludarabine: 30 mg/m2 over 30 minutes Day -6 through Day -2
  Busulfan: Busulfan 3.2 mg/kg IV once daily over 2-3 hours Day -4,-3,-2
Period: Overall Study
Arm/Group | CGD Recipient
Started | 7
Completed | 7 (Patient accrual was stopped early, and the protocol closed after completing followup)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CGD Recipient
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.42 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
  India | 1
Infection present [Count of Participants; unit: Participants] | 3
Autoimmunity present [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Efficacy of This Allogeneic Transplant Approach in Reconstituting Normal Hematopoiesis and Reversing the Clinical Phenotype of CGD
Description: Patient will have donor chimerism of greater than 20% and resolution of infection or autoimmunity at end of follow up
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | CGD Recipient
Number analyzed (Participants) | 7
Participants
  Greater than 20% donor chimerism | 7
  Resolution of inflammation or infection | 7

2. Secondary Outcome: To Determine the Safety of This Allogeneic HSCT Approach in Patients With CGD Including Transplant Related Toxicity, the Incidence of Acute and Chronic Graft-versus-host Disease, Immune Reconstitution, Overalland Disease-free Survival.
Description: 1. Stable chimerism as indicated by 30-50% myeloid engraftment and 50% lymphoid engraftment as assessed by 1 year post transplant. 2. Immune reconstitution levels with DHR as a marker of normal neutrophil function by 1 year post transplant. 3. GvHD grades of less than 3.
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | CGD Recipient
Number analyzed (Participants) | 7
Participants
  Number of patients with stable chimerism at 1 year | 6
  Patients with normal DHR at 1 year | 6
  Patients with Acute (Grade 3 or higher) GvHD | 3
  Patients with Chronic GvHD | 0
  Overall Survival | 5
  Disease Free Survival | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over 5 years (2015 to 2019)
Arm/Group | CGD Recipient
All-Cause Mortality (participants affected / at risk) | 2/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGD Recipient (N=7)
Severe Acute GvHD (Immune system disorders) | 3 (3)
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) — Development of irritation and bleeding from the bladder due to infection and/or chemotherapy
Post transplant lymphoproliferative disease (Blood and lymphatic system disorders) | 1 (1) — Development of a clonal outgrowth of cells due to suppression of the immune system
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGD Recipient (N=7)
Mild GvHD (Immune system disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT02282904/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT02282904/ICF_001.pdf